CLINICAL TRIAL: NCT01634503
Title: A Single Center, Open-label, Dose-escalating, Phase Ι Study to Evaluate the Safety of GX-188E Administered by Electroporation (EP) in DNA-based Therapeutic Vaccine for Patients With Cervical Intraepithelial Neoplasia Grade 3 (CIN 3)
Brief Title: Safety of GX-188E DNA Therapeutic Vaccine Administered by Electroporation to Cervical Intraepithelial Neoplasia Grade 3
Acronym: CIN3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GX-188E-SN
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Cervical Intraepithelial Neoplasia 3
Keywords: 3+3 design; Phase 1; Cervical Intraepithelial Neoplasia; Adult; Safety; Dose Finding
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1mg of GX-188E by electroporation (Experimental)
  Interventions: Genetic: GX-188E administered by electroporation
- 2mg of GX-188E by electroporation (Experimental)
  Interventions: Genetic: GX-188E administered by electroporation
- 4mg of GX-188E by electroporation (Experimental)
  Interventions: Genetic: GX-188E administered by electroporation

INTERVENTIONS:
Genetic: GX-188E administered by electroporation — Patients will be assigned to three dose groups:1mg, 2mg, and 4mg. Each patient will be administered GX-188E by electroporation in entire study period. The Maximum Tolerated Dose of GX-188E will be determined by the classical 3+3 dose escalation schedule. The number of patients will be ranged from 9 to 18.
  Other Names: Trigrid™ Delivery System

SUMMARY:
This study is to determine maximum tolerable dose (MTD) of GX 188E by defining the safety profile the safety and maximum tolerated dose of GX-188E administered by electroporation in Cervical Intraepithelial Neoplasia grade 3 (CIN 3) patients.

DETAILED DESCRIPTION:
This study is an open-label, dose-escalation, single-center, phase I study to evaluate the safety of GX-188E, a DNA-based therapeutic vaccine, administered by electroporation (EP) in patients with HPV-16 or HPV-18 associated cervical intraepithelial neoplasia grade 3 (CIN 3).

Each subject eligible to participate in the trial is given a subject number, which is assigned sequentially in ascending order, then allocated to only a single dose level of the drug. Three subjects are allocated at each dose level starting with 1mg whereby the dose is escalated in sequential subjects in ascending numerical order of subject ID.

Each subject visit the site three times for administration during the study and is given an intramuscular injection of GX-188E at a dose of 1mg, 2mg or 4mg by electroporation at each visit

The subjects conduct the follow-up visits twice, which are 8 weeks and 24 weeks after the third injection of GX-188E respectively.

ELIGIBILITY:
Inclusion Criteria:

* Female aged between 20 and 50(inclusive).
* Those who promised not to get pregnant from initiation to the first follow-up visit
* Who has diagnosed with Cervical Intraepithelial Neoplasia 3 by histopathologic examination and HPV type 16 or 18 detected
* Those who signed a voluntary written informed consent form for study participation.

Exclusion Criteria:

* Pregnant or lactating women.
* Administration of immunosuppressant or immunomodulator within 6 months prior to the enrollment
* Concomitant medication of any corticosteroid agents within 4 weeks prior to vaccination with the test drug
* Prior immunotherapy against HPV
* Administration of any blood products within 3 months prior to the screening visit
* Administration of any vaccine within 4 weeks prior to the screening visit (ex. Hepatitis A vaccine, Hepatitis B vaccine, Influenza vaccine, Td etc.)
* Positive serum test results for hepatitis C virus, hepatitis B virus surface antigen(HBsAg), or HIV
* Prior participation in any clinical trial within 30 days prior to the screening visit
* Patients predisposed to inflammatory reaction due to use of medical devices such as electroporation within 30 days of screening visit
* Past history of epilepsy or convulsion within 2 years prior to the screening visit
* At the discretion of the investigator, the skin condition covering deltoid muscles, within 2cm of the intended sites of injection, is not suitable for injection due to infection, ulcer, edema, tattoo, scar, injury etc.
* The thickness of skin fold covering deltoid muscles, intended injection sites, >40mm
* Any orthopedic artificial implant around the intended sites of electroporation (deltoid muscles)
* Any history of severe adverse drug events or severe allergic diseases
* Sinus bradycardia whose resting heart rate < 50beats/min.
* Pre-excitation syndrome such as Wolff-Parkinson-White syndrome
* Artificial implants or metallic implants
* Abnormal electrocardiography (ECG) including arrhythmia
* Any other ineligible condition at the discretion of the investigator that would be ineligible to participate the study

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2012-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Determination of maximum MTD by defining the safety profile of GX-188E | From baseline to end of study
  It would be determined based on the rate and severity grade of events or abnormalities through evaluating systemic or local adverse events, clinical laboratory test results, vital signs and so on.

SECONDARY OUTCOMES:
The expression levels of GX-188E in blood | At week -2, week 2, week 12 ,week 20 and week 36
Immunologic reactogenicity by measuring HPV E6 and E7 specific T cell response (IFN-γ ELISPOT) | At week -2, week 2, week 12 ,week 20 and week 36
The changes of the involved lesions and HPV infection status | Baseline, week 12 ,week 20 and week 36

CONTACTS AND LOCATIONS:
Overall Officials: Tae Jin Kim, Principal Investigator — Cheil General Hospital & Women's Healthcare Center
Locations (1):
- Cheil General Hospital & Women's Healthcare Center, Seoul, South Korea